CLINICAL TRIAL: NCT05066139
Title: Monocentric Randomized Study Evaluating the Impact of an Early Multidisciplinary Program in Elderly Subjects Starting a Chemotherapy for Digestive Cancer: Multidisciplinary Evaluation of Elderly Patients With Digestive Cancer (EPODIG-G)
Brief Title: Multidisciplinary Evaluation of Elderly Patients With Digestive Cancer (EPODIG-G)
Acronym: EPODIG-G
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Paul Strauss (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-018; 2021-A00956-35 (Other: [IDRCB])
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Digestive System Disease; Neoplasms
Keywords: Digestive cancer; supportive care; gastrointestinal cancer
MeSH Terms: conditions — Digestive System Diseases; Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A Standard of care (No Intervention): Patients will receive standard care before treatment initiation (i.e. geriatric assessment only).
  Geriatric assessment includes: Mini Mental State Examination ; mini-Geriatric Depression Scale (mini-GDS) ; Body Mass Index (BMI) calculation ; Mini Nutritional Assessment (MNA) ; Time up and Go ; Cumulative Illness Rating Scale - Geriatric (CIRS-G) ; Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL) questionnaires.
- Arm B Multidisciplinary EPODIG program (Experimental): Patients will undergo the same geriatric assessment as in Arm A plus EPODIG-G program before treatment initiation.
  Interventions: Other: EPODIG-G program (coordination of supportive care)

INTERVENTIONS:
Other: EPODIG-G program (coordination of supportive care) — EPODIG-G program includes: a nutritional evaluation (laboratory tests: albumin, pre-albumin, C reactive protein and vitamin D dosage, nutritional status, Handgrip test, Simple Evaluation of Food Intake (SEFI), spontaneous food intake evaluation) ; a medication reconciliation ; physical therapy (Six Minute Walk Test)
  Arms: Arm B Multidisciplinary EPODIG program

SUMMARY:
This is a monocentric, comparative, open-label, randomized parallel group study enrolling elderly subjects hospitalized in Strasbourg Europe Cancerology Institute (ICANS), starting chemotherapy or targeted therapy for the treatment of digestive cancer.

DETAILED DESCRIPTION:
At the ICANS an EPODIG-G program, consisting in a coordination of supportive care that are existing in the Institute, is proposed to elderly patients with digestive cancer. The purpose of this study is to evaluate the impact of this early multidisciplinary geriatric program (EPODIG-G), when it is initiated before therapeutic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 75 years old
* Performance status 0, 1 or 2
* Diagnostic of digestive cancer, all stages (adjuvant or metastatic), with an indication for chemotherapy treatment or targeted therapy for a treatment period of 24 weeks or more
* Patients previously treated with one or several lines of chemotherapy for this digestive cancer are eligible
* Estimated life expectancy ≥ 3 months
* Patients able to speak, read and understand French
* Signed informed consent from the patient
* Patients must have a social security coverage

Exclusion Criteria:

* History of differentiated neuroendocrine tumors grade 1 or 2 (pancreas, small intestine)
* Cancer currently being treated (except for hormone therapy) other than current digestive cancer
* History of major surgery and/or curative radiation therapy during the last 4 weeks before inclusion
* Patients unable to submit to medical follow-up for geographical, social or psychological reasons
* Patients placed under guardianship

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2030-10-17 (Estimated); Study Completion 2030-10-17 (Estimated)

PRIMARY OUTCOMES:
Impact of EPODIG-G program on treatment. | 24 weeks after treatment initiation
  Number of patients who benefit from all programmed treatment cycles at 24 weeks

SECONDARY OUTCOMES:
Dose-intensity evaluation. Cumulative doses and theoretical doses of chemotherapy or targeted therapy. | 24 weeks after treatment initiation
Number of adverse events and serious adverse events according to CTCAE v5.0. | throughout treatment, at 8, 16 and 24 weeks after treatment initiation
Progression free survival | 3 years after last inclusion
Overall survival | 3 years after last inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de cancérologie Strasbourg Europe, Strasbourg, France